CLINICAL TRIAL: NCT05961137
Title: Orange Park Out-of-Hospital Quality Improvement Study for Improving CMS Sepsis Core Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orange Park Medical Center (Other)
Collaborators: 410 Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1-1260269-1
Record Dates: First submitted 2023-05-22; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Sepsis; Emergency Medical Services; Quality Improvement; Shock, Septic; Fluid Therapy
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Intervention Model Description: Two-group design with control group enrolled first, then a training period, then a separate intervention group enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- After-phase: Incorporation of Rapid Fluid Infusion Device in Prehospital Suspected Sepsis Protocol (Active Comparator): Modified protocol specifying intravenous crystalloid infusion Rapid Fluid Infusion Device. The protocol states that for patients meeting the sepsis alert criterion, EMS will provide basic medical care, oxygen, a 12-lead electrocardiogram, attempt placement of an IV catheter and initiate administration of 30mL/kg of fluids.
  Interventions: Other: Incorporation of Rapid Fluid Infusion Device in Prehospital Suspected Sepsis Protocol
- Before phase: Conventional Prehospital Suspected Sepsis Protocol (Active Comparator): Conventional protocol employing intravenous crystalloid infusion via gravity or pressurized-bag. The protocol states that for patients meeting the sepsis alert criterion, EMS will provide basic medical care, oxygen, a 12-lead electrocardiogram, attempt placement of an IV catheter and initiate administration of 30mL/kg of fluids.
  Interventions: Other: Conventional Prehospital Suspected Sepsis Protocol

INTERVENTIONS:
Other: Incorporation of Rapid Fluid Infusion Device in Prehospital Suspected Sepsis Protocol — Modified protocol specifying intravenous crystalloid infusion Rapid Fluid Infusion Device. The protocol states that for patients meeting the sepsis alert criterion, EMS will provide basic medical care, oxygen, a 12-lead electrocardiogram, attempt placement of an IV catheter and initiate administration of 30mL/kg of fluids.
  Arms: After-phase: Incorporation of Rapid Fluid Infusion Device in Prehospital Suspected Sepsis Protocol
Other: Conventional Prehospital Suspected Sepsis Protocol — Conventional protocol employing intravenous crystalloid infusion via gravity or pressurized-bag. The protocol states that for patients meeting the sepsis alert criterion, EMS will provide basic medical care, oxygen, a 12-lead electrocardiogram, attempt placement of an IV catheter and initiate administration of 30mL/kg of fluids.
  Arms: Before phase: Conventional Prehospital Suspected Sepsis Protocol

SUMMARY:
The goal of this quality improvement study is to measure the impact of incorporation of a manual rapid fluid infuser (RFI) for intravenous crystalloid infusion in patients with suspected sepsis in the prehospital interval.

The main question[s] it aims to answer are:

* Does the intervention affect the timeliness of fluid administration?
* Does the intervention affect CMS sepsis bundle care measure compliance?
* Does the intervention affect processes and outcomes of care?
* Are there any adverse effects?

Researchers will compare this intervention to use of more conventional gravity or pressure-infusion bag crystalloid infusion.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting sepsis alert criteria who were transported to the study hospital's emergency department by one of the four rescue units involved in the study. Sepsis alert defined as patient has suspected infection and two or more of the following: (a) temperature > 38° C (100.4° F) or < 36° C (96.8° F), (b) respiratory rate > 20 breaths / minute or end-tidal carbon dioxide (ETCO2) ≤ 25 mmHg, or (c) heart rate > 90 beats / minute

Exclusion Criteria:

* prehospital trauma
* prehospital cardiac arrest prior to signaling sepsis alert
* interfacility transfer
* emergency transport from medical facility (e.g., medical office or clinic)
* intervention by medical practitioner before emergency medical services arrival
* do not resuscitate order in place

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Percentage compliance with the CMS 3-hour sepsis bundle criterion (SEP-1) for patients with suspected sepsis | Assessed at 3 hours after ED arrival
  As defined according to the Centers for Medicare and Medicaid Services (CMS) Specifications Manual for Hospital Inpatient Quality Measures, version 5.9. "Time of presentation" or "time-zero" was defined as the time of triage in the Emergency Department. All patients enrolled in the study were assessed for measure compliance, without application of measure inclusion/exclusion criteria.

SECONDARY OUTCOMES:
Percentage achievement of 30mL/kg crystalloid infusion for hypotension or lactate level > 4 mmol/L at 1 hour | Assessed at 1 hour after ED arrival
  Dichotomous measure of whether infusion volume was met, based on sum of prehospital and ED-based crystalloid fluid infusion
Total volume of intravenous crystalloid infused by time of ED arrival | During the 3 hours prior to ED arrival, while under care by EMS.
Total volume of intravenous crystalloid infused by 1 hour after ED arrival | Assessed at 1 hour after ED arrival
Total volume of intravenous crystalloid infused by 3 hours after ED arrival | Assessed at 3 hours after ED arrival
Total volume of intravenous crystalloid infused, in the ED, by 1 hour after ED arrival | Assessed at 1 hour after ED arrival
Total volume of intravenous crystalloid infused, in the ED, by 3 hours after ED arrival | Assessed at 3 hours after ED arrival
Percentage of study participants receiving any intensive care unit care | Through discharge from index acute-care episode, up to 6 months
Percentage of study participants with admission disposition during index ED visit | Through discharge from index acute-care episode, up to 6 months
Percentage of enrollees receiving any specified life-support interventions in the first 24 hours from ED arrival | Assessed at 24 hours after ED arrival
  Specified life-support interventions were mechanical ventilation, vasopressor use, cardiopulmonary resuscitation, surgical intervention.
Percentage of enrollees experiencing in-hospital death | Through discharge from index acute-care episode, up to 6 months
Total length of stay in ED | Through discharge from index acute-care episode, up to 6 months
  Operationalized as time difference between ED clinician's documented disposition time and the patient's arrival time.
Total length of stay in hospital | Through discharge from index acute-care episode, up to 6 months
  Among those admitted to the hospital as the disposition of their index ED visit.
Total length of stay in intensive care unit | Through discharge from index acute-care episode, up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin P Wegman, MD, PhD, Principal Investigator — Orange Park Medical Center
Locations (1):
- Orange Park Medical Center, Orange Park, Florida, United States

IPD SHARING:
Plan to Share IPD: No